CLINICAL TRIAL: NCT05124665
Title: Interrupting HIV and TB Stigma in the Household During TB Contact Investigation in Uganda
Brief Title: Interrupting HIV and TB Stigma in the Household in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); New York University (Other); Makerere University (Other); Walimu (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1R21TW011270 (NIH); 1R21TW011270-01 (NIH); 2000024852 (Other: Yale IRB)
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Hiv; Tuberculosis; Social Behavior; Stigma, Social; Stigmatization
Keywords: HIV; Tuberculosis; Stigma; Uganda
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Social Behavior; Social Stigma; Stereotyping | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: There are 3 teams of community health workers (CHWs) in total: one intervention, one standard of care, and one clinic-based that will always carry out initial enrollment and record clinic follow-up for both arms. Blinding of the CHWs is not feasible because it is a behavioral intervention that is easily recognized and CHWs must be trained to deliver either the standard of care or the intervention strategy. CHWs will collect data for the outcomes. CHWs will be separated into two teams and will only have electronic permissions to access training, procedures, forms, and contact information related to their assigned allocation within the electronic case record forms. They will be blinded to randomization procedures and outcomes. Participants will be blinded to their randomization assignment. Investigators and study staff will be blinded to study outcomes until the database is locked at the end of the trial. The onsite study coordinator who manages randomization will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Support (Experimental): CHWs will offer HIV testing to the individual nominated by the index patient as most likely to test. If this person is not present, CHWs will decide which contact should be offered testing first. CHWs will use a prosocial script for HIV testing: "Knowing your status sets a good example for your household." CHWs will follow an "opt-out" strategy: "This test kit is approved by the Ministry of Health and used in KCCA health facilities. I am going to offer you a free HIV test now, is that okay?". If the initial household contact who is offered HIV testing agrees to test, the CHW will ask if he/she is willing to share his/her decision to test with other members of the household: "Would you like to share your decision to test with the others? Sharing is completely optional. However, learning that someone else in their household decided to test sometimes gives people the strength to test themselves. Sharing your decision might help another person find the strength to test."
  Interventions: Behavioral: Social Support
- Standard of Care (No Intervention): As a control for the socio-behavioral intervention, the control arm will lack the socio-behavioral intervention components. The order of testing invitation will be decided by the CHW; and CHWs will be trained at baseline to provide standard, opt-in framing of test offers, without any mention of asking contacts to share their testing decision with other household contacts. Oral HIV kits will also be used in control households.

INTERVENTIONS:
Behavioral: Social Support — The intervention to be evaluated in this study is a multidimensional, socio-behavioral "Norming" intervention. The various components of this intervention are designed to harness household dynamics and prosocial inclinations to encourage individuals to accept the HIV testing invitation. Each component is briefly described in the arm description.
  Other Names: Intervention; Norming: Socio-Behavioral
  Arms: Social Support

SUMMARY:
The investigators will carry out a prospective, household cluster-randomized, implementation trial evaluating a complex, multi-component, social and behavioral intervention designed to normalize the acceptance of HIV testing in the household and increase diagnosis of HIV.

DETAILED DESCRIPTION:
An estimated 39 million people worldwide are living with HIV, but nearly half do not know their status because they are unaware that they are at risk, unable to access counseling and testing, or unwilling to accept testing because of stigma and fear. Layered on to the stigma of HIV is the risk of tuberculosis (TB), the leading cause of death among persons living with HIV (PLWH). Home testing is a promising approach to increase testing and linkage to care for HIV because it can reach individuals outside the health system, eliminate the costs of traveling for testing, offer testing in a familiar environment, and increase engagement with care among those found to be living with HIV. Nevertheless, many individuals offered home HIV testing in sub-Saharan Africa decline to test.

The investigators developed a complex intervention to increase uptake of testing for HIV among household members by reducing perceptions of stigma associated with HIV and testing for HIV. The intervention involves lay health workers (LHWs) delivering a novel invitation strategy for HIV testing in households that includes 1) acceptance-optimized sequencing, 2) prosocial messaging, and 3) salivary HIV testing. The investigators will administer HIV and TB stigma scales before and after the invitation. The investigators will conduct a household randomized controlled trial to test the intervention's impact on household HIV stigma and uptake of testing among household members undergoing TB contact investigation. The investigators will measure our co-primary outcomes of HIV and TB stigma using standardized instruments before invitation and after completion of post-test counseling. The investigators will measure the proportion consenting to HIV testing, yield of HIV diagnoses, and the proportion of new PLWH linked to HIV care at 1 month and reassess household HIV and TB stigma at 3 months.

This study will be conducted in Kampala, Uganda, and will involve TB index patients and their household contacts. Households will be recruited and enrolled through index patients initiating treatment for pulmonary tuberculosis (PTB) at Kampala Capital City Authority health facilities. The investigators will enroll index patients and their households from Kiswa, Kawaala, and Kisenyi Health Centers, each a public-sector, primary care facility.

This study will enroll households (index patients + their household contacts). Only household contacts are eligible for participation; close contacts are not eligible. For the purposes of this study, household contacts are defined as those individuals "sleeping under the same roof" as the index patient for one or more nights within the past three months.

Upon encountering a patient initiating treatment for TB or returning for 2-week follow-up, study CHWs will assess index patients for household-level eligibility for the study. All index patients whose households meet these criteria will be asked to provide verbal consent after reviewing an information sheet. If the index patient is a minor (age < 18 years), the guardian of the index patient will be asked to provide verbal consent.

After study enrollment, a CHW will work with the index patient and, if available, treatment supporter to schedule the home visit. Households will be randomly assigned to one of the two CHW teams to receive the intervention or standard or care strategy.

After the enrollment of the household through the index patient, household contact investigation will take place. All household contacts who meet these criteria will be asked to provide verbal consent after reviewing an information sheet. If the contact is a minor (aged 15-17), he or she will be asked to provide verbal assent with his/her parent/guardian providing consent. Enrolling in the study does not require eligibility for or consent to HIV testing. Those who choose to participate in the study and are eligible for HIV testing will be subsequently offered testing and may consent or decline. Those who choose to participate in the study and report conditions that render them ineligible for HIV testing, such as already known to be a PLWH, testing negative within the last three months, or currently in TB treatment, will not be offered HIV testing but will be eligible to participate in other study procedures.

Variable block randomization will be done at the level of the household and will be performed at the time of household enrollment. Block sizes will have a minimum of 4 households, a maximum of 8 households. The investigators will utilize Study Randomizer, an online randomization tool with concealed allocation, to generate the allocation sequence. When a CHW determines that an index patient is eligible for the study, and after the index patient or guardian has provided verbal informed consent, the CHW will place a phone call to the study coordinator. The study coordinator will then enroll the household using the Study Randomizer tool and let the CHW know the study allocation. The CHW will then record the appropriate allocation in the survey software, along with the randomization ID, and contact the appropriate CHW team for the household visit. The index patient will be given the name of the community health worker who will be visiting the household, and immediately connected with that person by telephone to arrange the home visit.

Households randomized to intervention group (Social Support Group) will be offered the social-behavioral intervention. Households randomized to the standard of care group (Standard of Care) will be offered oral testing without any social-behavioral intervention. CHWs will operate in teams that are always assigned to the same arm of the study. There will be three teams of CHWs in total: one intervention group, one standard of care group, and one clinic-based group that will always carry out initial enrollment of index patients and record any clinic follow-up by individuals in either arm of the study.

Regardless of intervention or control arm, CHWs will deliver a short, 13-item TB and HIV stigma scale to all household contacts at the beginning (prior to TB evaluation) and end of the household visit (after all TB and HIV procedures). The scale was adapted from the Van Rie TB HIV stigma scale specifically for this context. The scales will be administered first at the beginning of the home visit, then again at its conclusion.

The primary outcome is uptake of HIV testing, defined as the proportion of eligible individuals in the household who undergo testing after a test offer compared between the intervention arm and the standard of care arm..

ELIGIBILITY:
Index Patient and Household Eligibility:

* Index patient is eligible for contact investigation (TB patient of any age identified in the facility's National TB and Leprosy Programme (NTLP) TB Treatment Register as initiating treatment or returning for 2-week follow-up)
* Index patient or legal guardian agrees to study procedures in addition to routine contact investigation
* Index patient has at least 2 self-reported household contacts age 15 or above
* Household is within the boundaries of the Kampala Capital City Authority, Uganda
* Does not have multi-drug resistant (MDR) TB

Contact Participant Eligibility:

* Household contact age ≥15 years
* Agrees to study procedures in addition to routine contact investigation

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Lucian Davis, MD, Principal Investigator — Yale School of Public Health; Achilles Katamba, PhD, Principal Investigator — Makerere University; Mari Armstrong-Hough, PhD, Principal Investigator — New York University
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified will be available upon request after the publication of main trial results. Individuals interested in data must reach out to one of the principal investigators.
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of main trial results. Data will be held by the researchers for a minimum of 7 years after the end of the trial.
Access Criteria: A research proposal must be submitted to one of the principal investigators outlining the type of data needed as well as intended use of data.

REFERENCES:
- [Background] Armstrong-Hough M, Ggita J, Gupta AJ, Shelby T, Nangendo J, Ayen DO, Davis JL, Katamba A. Assessing a norming intervention to promote acceptance of HIV testing and reduce stigma during household tuberculosis contact investigation: protocol for a cluster-randomised trial. BMJ Open. 2022 May 25;12(5):e061508. doi: 10.1136/bmjopen-2022-061508. PMID 35613785
- [Derived] Armstrong-Hough M, Gupta AJ, Ggita J, Nangendo J, Katamba A, Davis JL. Using group norms to promote acceptance of HIV testing during household tuberculosis contact investigation: A household-randomized trial. medRxiv [Preprint]. 2024 May 3:2024.05.02.24306703. doi: 10.1101/2024.05.02.24306703. PMID 38746428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 208 index participants were randomized to be contacted for either Social Support or Standard of Care were identified and randomized to be approached in the community. Presented are the totals that agreed to participate in terms of the number of index participants that consented to participants and then added household contacts that consented to also participate.
Period: Overall Study
Arm/Group | Social Support | Standard of Care
Started (Index participants randomized that agreed to participate in the study and then the household contacts that agreed to participate.) | 364 | 248
Index Patients | 79 | 61
Household Contacts | 285 | 187
Completed | 364 | 248
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Provided are baseline characteristics for all that participated- both index and household contact participants.
Groups:
- Social Support: Household Contacts: CHWs will offer HIV testing to the individual nominated by the index patient as most likely to test. If this person is not present, CHWs will decide which contact should be offered testing first. CHWs will use a prosocial script for HIV testing: "Knowing your status sets a good example for your household." CHWs will follow an "opt-out" strategy: "This test kit is approved by the Ministry of Health and used in KCCA health facilities. I am going to offer you a free HIV test now, is that okay?". If the initial household contact who is offered HIV testing agrees to test, the CHW will ask if he/she is willing to share his/her decision to test with other members of the household: "Would you like to share your decision to test with the others? Sharing is completely optional. However, learning that someone else in their household decided to test sometimes gives people the strength to test themselves. Sharing your decision might help another person find the strength to test."
  Social Support: The intervention to be evaluated in this study is a multidimensional, socio-behavioral "Norming" intervention. The various components of this intervention are designed to harness household dynamics and prosocial inclinations to encourage individuals to accept the HIV testing invitation. Each component is briefly described in the arm description.
- Social Support: Index Participants: Social Support: The intervention to be evaluated in this study is a multidimensional, socio-behavioral "Norming" intervention. The various components of this intervention are designed to harness household dynamics and prosocial inclinations to encourage individuals to accept the HIV testing invitation. Each component is briefly described in the arm description.
- Standard of Care: Household Contacts; Standard of Care: Index Participants: As a control for the socio-behavioral intervention, the control arm will lack the socio-behavioral intervention components. The order of testing invitation will be decided by the CHW; and CHWs will be trained at baseline to provide standard, opt-in framing of test offers, without any mention of asking contacts to share their testing decision with other household contacts. Oral HIV kits will also be used in control households.
- Total: Total of all reporting groups
Arm/Group | Social Support: Household Contacts | Social Support: Index Participants | Standard of Care: Household Contacts | Standard of Care: Index Participants | Total
Number analyzed (Participants) | 285 | 79 | 187 | 61 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (12.7) | 31.3 (16.9) | 31.4 (14.4) | 28.6 (18.5) | 30.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 35 | 122 | 22 | 366
  Male | 98 | 44 | 65 | 39 | 246
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Count of Index Participants
  participants
    Uganda | 285 | 79 | 187 | 61 | 612
HIV Status [Count of Participants; unit: Participants]
  Not Known to be Living with HIV | 224 | 50 | 152 | 49 | 475
  Unknown/Never Tested | 61 | 0 | 35 | 0 | 96
  Person Living with HIV | 0 | 29 | 0 | 12 | 41
Education Level [Count of Participants; unit: Participants] — Population: Education data collected only for Household Contacts
  Participants
    number analyzed (Participants) | 285 | 0 | 187 | 0 | 472
    No Formal Education | 13 |  | 7 |  | 20
    Level 1-4 | 22 |  | 15 |  | 37
    Level 5-7 | 66 |  | 50 |  | 116
    O-Level | 104 |  | 66 |  | 170
    A-Level | 38 |  | 18 |  | 56
    Vocational | 5 |  | 5 |  | 10
    Tertiary/University | 31 |  | 24 |  | 55
    Post-Graduate | 6 |  | 2 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Contacts Accepting HIV Testing
Description: To test the hypothesis that a norming intervention can increase test uptake, the investigators will compare testing uptake among the intervention households and control households using cluster-adjusted chi-squared tests of proportion and by fitting mixed effects logistic regression models with two levels (household, contact). The effect of the intervention will then be evaluated by comparing adjusted slope differences in the primary outcomes (test uptake) between the intervention and the control arms, using random intercept mixed logit models to account for clustering by household.
Time Frame: up to 8 weeks
Population: Household Contacts
Measure: Count of Participants; unit: Participants
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 285 | 187
Participants | 279 | 172
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is that proportion of contacts accepting HIV testing between two study arms is equivalent; p = 0.004, Mixed Models Analysis; Cluster adjusted for household; Odds Ratio (OR) = 4.6, 95% CI 2-sided [1.6 to 12.9]
Statistical Analysis 2: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is proportion of contacts accepting HIV testing is equivalent between the two study arms; p = 0.006, t-test, 2 sided; Mean Difference (Net) = 6, 95% CI 2-sided [2 to 10] — Estimated value and confidence interval reflects the values multiplied by 100 (converting decimal to percentage)

2. Secondary Outcome: Change in Score of Perceived HIV Stigma
Description: Change in HIV Stigma will be evaluated by measuring the change in HIV-TB stigma as measured by the Van Rie paired HIV-TB Stigma Scales (adapted for use in Uganda) using multilevel models. The investigators will use mixed effects Poisson regression models to evaluate changes in HIV stigma measured after the household visit among a two-stage,stratified random sample of participants.
  Van Rie Perceived TB and HIV Stigma scales adapted and validated in the Ugandan context are used. Scores range from 0 to 100 (standardized scale). Higher values represent higher levels of perceived stigma. The timeframe has been updated to reflect changes in follow up due to COVID-19 restrictions.
Time Frame: Baseline to End of Interview (Up to 8 hours)
Population: Household Contacts
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 285 | 187
score on a scale | 2.57 (24.9) | -0.21 (18.6)
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Van Rie Perceived TB and HIV Stigma scales adapted and validated in the Ugandan context are used. Scores range from 0 to 100 (standardized scale); Test type: Equivalence — Hypothesis is that the change in stigma score is equivalent between the two study arms; p = 0.358, Mixed Models Analysis; Slope = 2.20, 95% CI 2-sided [-2.5 to 6.9]

3. Secondary Outcome: Change in Score of Perceived TB Stigma
Description: Change in TB Stigma will be evaluated by measuring the change in perceived TB stigma as measured by the Van Rie paired HIV-TB Stigma Scales (adapted for use in Uganda) using multilevel models. The investigators will use mixed effects Poisson regression models to evaluate changes in TB stigma measured after the household visit among a two-stage,stratified random sample of participants.
  Van Rie Perceived TB and HIV Stigma scales adapted and validated in the Ugandan context are used. Scores range from 0 to 100 (standardized scale). Higher values represent higher levels of perceived stigma. The timeframe has been updated to reflect changes in follow up due to COVID-19 restrictions.
Time Frame: Baseline to End of Interview (Up to 8 hours)
Population: Household Contacts
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 285 | 187
score on a scale | 0.47 (20.8) | -2.52 (17.8)
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is that the difference in stigma score is equivalent between the two study arms; p = 0.199, Mixed Models Analysis; Slope = 2.61, 95% CI 2-sided [-1.38 to 6.59]

4. Secondary Outcome: Change in Effects of Perceived HIV Stigma on HIV Test Uptake
Description: The investigators will conduct a causal mediation analysis to determine the degree to which the effects of the intervention on HIV stigma explain the improvement in HIV test uptake using observed-variable structural equation modeling. HIV stigma will be measured using the Van Rie paired HIV-TB Stigma Scales (adapted for use in Uganda) and standardized scores (0 to 100) will be utilized. Higher score represents higher levels of perceived stigma.
Time Frame: Baseline to Immediately post intervention (up to 8 hours)
Population: Household Contacts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 285 | 187
units on a scale | 2.59 (24.75) | -0.17 (20.09)
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is no effect from perceived HIV Stigma on HIV Test Uptake; p = 0.03, Structural Equation Modeling; Coefficient from Structural Equation = 0.00087, 95% CI 2-sided [0.00007 to 0.00167]

5. Secondary Outcome: Change in Effects of Perceived TB Stigma on HIV Test Uptake
Description: The investigators will conduct a causal mediation analysis to determine the degree to which the effects of the intervention on TB stigma explain the improvement in HIV test uptake using observed-variable structural equation modeling. TB stigma will be measured using the Van Rie paired HIV-TB Stigma Scales (adapted for use in Uganda) and standardized scores (0 to 100) will be utilized. Higher score represents higher levels of perceived stigma.
Time Frame: Baseline to End of Interview (Up to 8 hours)
Population: Household Contacts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 285 | 187
units on a scale | -0.46 (21.12) | -2.34 (16.82)
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is that TB stigma has no effect of HIV test uptake; p = 0.64, Structural Equation Modeling; Coefficient Structural Equation Model = 0.0002, 95% CI 2-sided [-0.0007 to 0.0011]

6. Secondary Outcome: Proportion of Index Patient Nominated Household Members Who Accept HIV Test
Description: The investigators will measure the proportion of testing preference predictions made by the index patient about their household contacts that were accurate, that is, the proportion of household members who accepted the HIV test among those nominated by the index patient as being most likely to accept the HIV test. The proportion of first testers who accepted the HIV test in the intervention arm will be compared to the proportion of first testers who took the HIV test in the control arm.
Time Frame: up to 8 weeks
Population: Household Contacts
Measure: Count of Participants; unit: Participants
Groups:
- Social Support: Household Contacts: Individuals nominated to be the first HIV tester in the household within the Social Support Arm
- Standard of Care: Household Contacts: Individuals nominated to be the first HIV tester in the household within the Standard of Care Arm
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 59 | 33
Participants | 58 | 33
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is that proportion of index patient nominated household contacts accepting HIV testing is equivalent between two study arms; p = 0.452, Chi-squared

7. Secondary Outcome: Number of Social Support Household Contacts Deciding to Test for HIV
Description: The investigators will estimate in the intervention arm the effect of first testers' decision to disclose on subsequent testers' decisions to test in the intervention arm using a logistic regression model. This will be assessed with relative risk of first testers' decision to disclose testing decision on subsequent household members decision to test for HIV.
Time Frame: up to 8 weeks
Population: Household Contacts
Measure: Count of Participants; unit: Participants
Groups:
- Social Support: Household Contacts: Individuals who were NOT the first person asked to test for HIV in the household within the Social Support Arm of the trial. This is to understand the impact of the first tester's decision to test on subsequent testing decisions. Therefore, only those who were NOT offered HIV testing first in the Social Support arm of the trial are included.
Arm/Group | Social Support: Household Contacts
Number analyzed (Participants) | 285
Participants | 196
Statistical Analysis 1: Comparison: Social Support: Household Contacts; Test type: Non-Inferiority — Hypothesis is that the first tester's decision to test does not impact subsequent household contacts decision to test for HIV; p = 0.264, Regression, Logistic; Risk Ratio (RR) = 1.23, 95% CI 2-sided [0.86 to 1.76]

8. Other Pre Specified Outcome: Count of Social Influence Nominations (Participants) by the Index Patient That Align With Nominations by the Household Contacts
Description: The investigators will assess the concordance of index patients' perceptions of their household contacts' influence on health decisions within the household with the perceptions of the rest of their household. To do so, the investigators will measure the number of participants that provide social influence nominations that align with nominations by the household contacts in the intervention arm.
Time Frame: up to 8 weeks
Population: Only includes contacts who provided a nomination for social influence within the household (subset of all household contacts)
Measure: Count of Participants; unit: Participants
Groups:
- Social Support: Household Contacts: Household contacts who provided a nomination for social influence within the household (subset of all contacts) for the social support arm
- Standard of Care: Household Contacts: Household contacts who provided a nomination for social influence within the household (subset of all contacts) for the standard of care arm
Arm/Group | Social Support: Household Contacts | Standard of Care: Household Contacts
Number analyzed (Participants) | 246 | 152
Participants | 148 | 59
Statistical Analysis 1: Comparison: Social Support: Household Contacts vs Standard of Care: Household Contacts; Test type: Equivalence — Hypothesis is that the index patient and contact nominations will match equally regardless of study arm; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 3 months post intervention delivery
Description: Adverse events were collected on all participants- including index participants and household contacts.
Groups:
- Social Support: Index Participants; Social Support: Household Contacts: CHWs will offer HIV testing to the individual nominated by the index patient as most likely to test. If this person is not present, CHWs will decide which contact should be offered testing first. CHWs will use a prosocial script for HIV testing: "Knowing your status sets a good example for your household." CHWs will follow an "opt-out" strategy: "This test kit is approved by the Ministry of Health and used in KCCA health facilities. I am going to offer you a free HIV test now, is that okay?". If the initial household contact who is offered HIV testing agrees to test, the CHW will ask if he/she is willing to share his/her decision to test with other members of the household: "Would you like to share your decision to test with the others? Sharing is completely optional. However, learning that someone else in their household decided to test sometimes gives people the strength to test themselves. Sharing your decision might help another person find the strength to test."
  Social Support: The intervention to be evaluated in this study is a multidimensional, socio-behavioral "Norming" intervention. The various components of this intervention are designed to harness household dynamics and prosocial inclinations to encourage individuals to accept the HIV testing invitation. Each component is briefly described in the arm description.
Arm/Group | Social Support: Index Participants | Social Support: Household Contacts | Standard of Care: Index Participants | Standard of Care: Household Contacts
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/285 | 0/61 | 0/187
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/285 | 0/61 | 0/187
Other Adverse Events (participants affected / at risk) | 0/79 | 0/285 | 0/61 | 0/187

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT05124665/Prot_SAP_002.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT05124665/ICF_001.pdf